CLINICAL TRIAL: NCT00662844
Title: Optimum Vitamin D Nutrition in Young Women
Brief Title: Vitamin D Supplementation in Younger Women
Acronym: VITADAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PR065013; DOD. CDMRP. W81XWH-07-1-0201 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Hypovitaminosis D
Keywords: Vitamin D insufficiency,vitamin D3 treatment,young women
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Calcium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A1 vitamin D3 400IU (Placebo Comparator): Orally for one year
  Interventions: Dietary Supplement: vitamin D3
- A2 vitamin D3 800IU (Placebo Comparator): Orally for one year
  Interventions: Dietary Supplement: vitamin D3
- A3 vitamin D3 1600IU (Placebo Comparator): Orally for one year
  Interventions: Dietary Supplement: vitamin D3
- A4 Vitamin D3 2400 IU (Placebo Comparator): Orally for one year
  Interventions: Dietary Supplement: vitamin D3
- Placebo (Placebo Comparator): Placebo for one year
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Oral, one capsule daily of vitamin D3 (400IU, 800IU, 1600 IU, or 2400IU) plus calcium citrate (1-4 tablets) twice daily to reach a total calcium intake of 1000-1200 mg/day
  Other Names: Calcium citrate (Citracal)

SUMMARY:
That on average it will require a vitamin D dose of 1700IU/day to increase the serum 25hydroxyvitamin D level from 20 to 30ng/ml in young Caucasian women and a dose of 1860 to 2480 IU/day in African American

DETAILED DESCRIPTION:
Vitamin D is a unique nutrient in that its requirement can be met by both endogenous production from sun and from diet, which makes it difficult to determine the actual requirements as for other nutrients. The current recommended dietary reference intake (DRI) for vitamin D is 200 IU for adults between 25- 50 years, 400 IU for adults between 51-70 years and 600 IU for adults 70 years of age. In view of many scientists in the field of vitamin D, the current DRI of vitamin D is too low. This is mainly because of the increase in prevalence of vitamin D deficiency observed in the population based on measured serum 25OHD levels. It is now recognized that serum 25OHD is an indicator of vitamin D status. There is a growing consensus that serum 25OHD concentration of at least 30-32 ng/ml are needed to reduce serum Parathyroid hormone (PTH) and reduce bone loss. Also, research over the last two decades has provided additional evidence that higher vitamin D levels (25OHD 30ng/ml) are necessary for optimum overall health and prevent disease. There is no clear view of the amount of vitamin D intake required to maintain the optimum level of serum 25OHD levels in the population of all ages and there are no systematic dose response studies of vitamin D in women of all ages. A few studies carried out with different sexes and age groups have suggested that an untreated subject with a serum 25OHD concentration of 20 ng/ml would need a daily dose of ~1700 IU/d of Vitamin D3 to reach a serum 25OHD of 32 ng/ml in Caucasians, while in African Americans the Vitamin D3 requirement would be higher - 1860-2480 IU/d.

The current proposal aims at studying the dose response effect of vitamin D3 400 IU, 800 IU,1600 IU and 2400 IU or placebo on serum 25OHD and serum PTH in young women with vitamin D insufficiency (serum 25OHD <20 ng/ml) and an adequate calcium intake of 1000mg/day.

Another aim of the study is to establish the minimum effective dose of vitamin D3 which Normalizes PTH in Caucasian and African American young women. Vitamin D dose that reduces serum PTH to normal level in 97% of normal population is the recommended dietary allowance.

We will also establish the safety of these higher doses of vitamin D supplementation relating to hypercalcemia/hypercalcuria.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women, minimum age 25 years, maximum age 45 years. (Women with hysterectomy and/or oophorectomy must have a premenopausal FSH level.)
2. Serum 25OHD level: 5 - 20 ng/ml
3. BMI < 45 kg/m2.
4. Willing to discontinue vitamin D supplements after entering the study.
5. Negative pregnancy test before BMD and calcium absorption tests.
6. Willing to give signed informed consent form
7. Subject is Caucasian or African American

Exclusion Criteria:

1. Cancer (exceptions: basal cell carcinoma or if cancer occurred more than 10 years ago) or terminal illness.
2. Previous hip fracture.
3. Hemiplegia.
4. Uncontrolled type I diabetes ± significant proteinuria or fasting blood sugar >140 mg in type II diabetes.
5. Kidney stones- > 2 in a lifetime.
6. Chronic renal failure (serum creatinine >1.4 mg/dl).
7. Evidence of chronic liver disease, including alcoholism.
8. Physical conditions such as severe osteoarthritis, rheumatoid arthritis, heart failure severe enough to prevent reasonable physical activity.
9. Previous treatment with bisphosphonates (more that 3 months), PTH or PTH derivatives, (e.g. Teriparatide) or Fluoride in the last 6 months.
10. Previous treatment within the last 6 months with calcitonin or estrogen (except birth control pills).
11. Chronic high dose corticosteroid therapy (> 10 mg/day) for over 6 months and not within the last 6 months.
12. Anticonvulsant therapy. (Dilantin, Phenobarbital)
13. High dose thiazide therapy (> 37.5 mg).
14. 24 hour urine calcium > 290 mg on 2 baseline tests.
15. Serum calcium exceeding upper normal limit on 2 baseline tests.
16. BMD. T-score less than -3.0 for spine or hip.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2008-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Serum 25hydroxyvitamin D | Baseline, Change from Baseline at 6 Months and 12 Months
Parathyroid hormone | Baseline, Change from Baseline at 6 Months and 12 Months

SECONDARY OUTCOMES:
serum and urine calcium | Baseline, Change from Baseline at 6 Months, 9 Months and 12 Months
calcium absorption | Baseline, Change from Baseline at 12 Months
  radioactive calcium absorption is measured at baseline and end of study
Bone density | Baseline, Change from Baseline at 12 Months
  bone density
physical performance battery | Baseline, Change from Baseline at 12 Months
Forced Expiratory Volume FEV1 | Baseline, Change from Baseline at 12 Months
  spirometry
bone markers | Baseline, Change from Baseline at 12 Months
  serum osteocalcin,serum N-telopeptides
Serum 1,25-dihydroxyvitamin D3 | Baseline, Change from Baseline at 12 Months
  serum test
skin color | Baseline, Change from Baseline at 6 Months and 12 Months
  measurement of sin color through the study using an IMS smart probe
Serum 24,25dihydroxyvitamin D | Baseline, Change from Baseline at 12 Months
  measurement of serum 24,24(OH)2D by LCMS( liquid chromatography mass spectrophotometry

CONTACTS AND LOCATIONS:
Overall Officials: J C Gallagher, MD, Principal Investigator — Creighton University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallagher JC, Kinyamu HK, Fowler SE, Dawson-Hughes B, Dalsky GP, Sherman SS. Calciotropic hormones and bone markers in the elderly. J Bone Miner Res. 1998 Mar;13(3):475-82. doi: 10.1359/jbmr.1998.13.3.475. PMID 9525348
- [Background] Aloia JF, Talwar SA, Pollack S, Feuerman M, Yeh JK. Optimal vitamin D status and serum parathyroid hormone concentrations in African American women. Am J Clin Nutr. 2006 Sep;84(3):602-9. doi: 10.1093/ajcn/84.3.602. PMID 16960175
- [Background] Holick MF, Siris ES, Binkley N, Beard MK, Khan A, Katzer JT, Petruschke RA, Chen E, de Papp AE. Prevalence of Vitamin D inadequacy among postmenopausal North American women receiving osteoporosis therapy. J Clin Endocrinol Metab. 2005 Jun;90(6):3215-24. doi: 10.1210/jc.2004-2364. Epub 2005 Mar 29. PMID 15797954